CLINICAL TRIAL: NCT01954550
Title: Aerobic Exercise in Alzheimer's Disease: Cognition and Hippocampal Volume Effects
Brief Title: Effects of Aerobic Exercise for Treating Alzheimer's Disease
Acronym: FIT-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Mayo Clinic (Other); University of St Thomas (Unknown); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1306M356; 1R01AG043392-01A1 (NIH)
Record Dates: First submitted 2013-09-20; First posted 2013-10-01 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Alzheimer's Disease, Late Onset
Keywords: Exercise; Dementia; Cognition; Brain Volume; Aging
MeSH Terms: conditions — Alzheimer Disease; Motor Activity; Dementia | interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cycling exercise (Experimental): An exercise interventionist will guide and supervise participants to participate in moderate-intensity cycling on recumbent stationary cycles for 20-50 minutes, 3 times a week for 6 months.
  Interventions: Behavioral: Cycling exercise
- Range of motion/stretching exercise (Sham Comparator): An exercise interventionist will guide and supervise participants to participate in low-intensity range of motion/stretching exercise for 20-50 minutes, 3 times a week for 6 months.
  Interventions: Behavioral: Range of motion/stretching exercise

INTERVENTIONS:
Behavioral: Cycling exercise — An exercise interventionist will guide and supervise participants to participate in moderate-intensity cycling on recumbent stationary cycles for 20-50 minutes, 3 times a week for 6 months.
  Arms: Cycling exercise
Behavioral: Range of motion/stretching exercise — An exercise interventionist will guide and supervise participants to participate in low-intensity range of motion/stretching exercise for 20-50 minutes, 3 times a week for 6 months.
  Arms: Range of motion/stretching exercise

SUMMARY:
This randomized controlled trial (RCT) will investigate the effects of a 6-month, individualized, moderate-intensity cycling intervention on cognition and hippocampal volume in AD with three aims:

* Determine the immediate effect of the cycling intervention on cognition in AD.
* Examine if the cycling intervention slows cognitive decline in AD from baseline to 12 months.
* Assess the effect of aerobic exercise on hippocampal volume in AD over 12 months using MRI.

The investigators will randomize 90 participants to the 6-month cycling or stretching/range of motion exercise (20-50-minute, 3 times a week). Participants will then be followed for another 6 months. Cognition will be assessed at baseline, 3, 6, 9, and 12 months and hippocampal volume will be measured using magnetic resonance imaging (MRI) at baseline, 6, and 12 months.

DETAILED DESCRIPTION:
Aerobic exercise holds great promise for treating cognitive impairment, the hallmark symptom of Alzheimer's disease (AD), because it may attenuate brain atrophy. AD currently affects more than 5 million Americans, costing $203 billion in 2013 and causing poor outcomes such as loss of independence, low quality of life, and nursing home placement. Available drugs have only modest short-term effects on reducing or slowing cognitive impairment in AD. Hence, there is a pressing need to develop and test aerobic exercise interventions for AD. This randomized controlled trial (RCT) will investigate the effects of a 6-month, individualized, moderate-intensity cycling intervention on cognition and hippocampal volume in AD with three aims:

* Determine the immediate effect of the cycling intervention on cognition in AD.
* Examine if the cycling intervention slows cognitive decline in AD from baseline to 12 months.
* Assess the effect of aerobic exercise on hippocampal volume in AD over 12 months using MRI.

The investigators will randomize 90 participants to the 6-month cycling or stretching/range of motion exercise (20-50-minute, 3 times a week). Participants will then be followed for another 6 months. Cognition will be assessed at baseline, 3, 6, 9, and 12 months and hippocampal volume will be measured using magnetic resonance imaging (MRI) at baseline, 6, and 12 months. Transportation will be provided to participants for all study-related activities including exercises. Participants who could not undergo MRI can still participate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or possible Alzheimer's disease (AD);
* 15≤ Mini-Mental State Examination (MMSE) score ≤26;
* Clinical Dementia Rating score 0.5-2;
* Community-dwelling, e.g., homes and assisted living;
* Age 66 years and older;
* English-speaking;
* Verified exercise safety by the primary care providers and the cardiologists if subjects have significant cardiac history;
* Stable on AD drugs >1 month if AD drugs are prescribed.

Exclusion Criteria:

* Resting heart rate (HR) ≤50 or ≥100 beats/min;
* Neurological disorders in the past 5 years;
* Psychiatric disorders in the past 5 years;
* Alcohol or chemical dependency in the past 5 years;
* Contraindications to exercise;
* New symptoms or diseases that have not been evaluated by a health care provider, e.g., hip fracture, ongoing and unplanned weight loss, severe shortness of breath, deep vein thrombosis, hernia, unhealed sores, joint swelling, pain or trouble walking;
* Cardiac ischemia or serious arrhythmia on the electrocardiograph during the screening exercise test.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in cognition from baseline to 6 months as measured by the Alzheimer's Disease Assessment Scale - Cognitive Subscale | Baseline, 3 months, 6 months, 9 months, and 12 months
  This outcome measure will be given to all study participants.

SECONDARY OUTCOMES:
Change in hippocampal volume as measured by Magnetic Resonance Imaging (MRI) | Baseline, 6 months, and 12 months
  Only participants who qualified to undergo MRI will be assessed for hippocampal volume.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yu, PhD, Principal Investigator — Nursing
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu F, Bronas UG, Konety S, Nelson NW, Dysken M, Jack C Jr, Wyman JF, Vock D, Smith G. Effects of aerobic exercise on cognition and hippocampal volume in Alzheimer's disease: study protocol of a randomized controlled trial (The FIT-AD trial). Trials. 2014 Oct 11;15:394. doi: 10.1186/1745-6215-15-394. PMID 25304364
- [Derived] Yu F, Han SY, Salisbury D, Pruzin JJ, Geda Y, Caselli RJ, Li D. Feasibility and preliminary effects of exercise interventions on plasma biomarkers of Alzheimer's disease in the FIT-AD trial: a randomized pilot study in older adults with Alzheimer's dementia. Pilot Feasibility Stud. 2022 Dec 2;8(1):243. doi: 10.1186/s40814-022-01200-2. PMID 36461134
- [Derived] Yu F, Mathiason MA, Han S, Gunter JL, Jones D, Botha H, Jack C Jr. Mechanistic Effects of Aerobic Exercise in Alzheimer's Disease: Imaging Findings From the Pilot FIT-AD Trial. Front Aging Neurosci. 2021 Oct 7;13:703691. doi: 10.3389/fnagi.2021.703691. eCollection 2021. PMID 34690736
- [Derived] Greimel S, Wyman JF, Zhang L, Yu F. Recruitment and Screening Methods in Alzheimer's Disease Research: The FIT-AD Trial. J Gerontol A Biol Sci Med Sci. 2022 Mar 3;77(3):547-553. doi: 10.1093/gerona/glab092. PMID 33780529
- [Derived] Li D, Thomas R, Tsai MY, Li L, Vock DM, Greimel S, Yu F. Vascular biomarkers to predict response to exercise in Alzheimer's disease: the study protocol. BMJ Open. 2016 Dec 30;6(12):e011054. doi: 10.1136/bmjopen-2016-011054. PMID 28039287
- See also: Study Listing at the Alzheimer's Association — https://trialmatch.alz.org/trialsearch/Public/TrialSummary.aspx?trialID=78871&diseaseID=1626&subdiseaseID=1666&i_user_type=physician